CLINICAL TRIAL: NCT06627283
Title: Effects of Respiratory Muscle Training on Tongue Muscle Function in Healthy Subjects, a Randomized Controlled Trial.
Brief Title: Effects of Respiratory Muscle Training on Tongue Muscle Function
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Université Catholique de Louvain (Other)
Responsible Party: Principal Investigator, William Poncin, PhD, Université Catholique de Louvain
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: RMT-TONGUE
Record Dates: First submitted 2024-10-02; First posted 2024-10-04 (Actual); Last update posted 2024-12-10 (Actual); Status verified 2024-12

CONDITIONS: Healthy

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- IMT (Active Comparator)
  Interventions: Device: IMT
- EMT (Active Comparator)
  Interventions: Device: EMT
- Sham (Sham Comparator)
  Interventions: Device: Sham
- Control (No Intervention)

INTERVENTIONS:
Device: IMT — Description: A pressure threshold loading device will be used: the POWERbreathe Medic (load range 10-90 cmH2O). Participants will be instructed to exhale passively during normal tidal breathing through the training device (until functional residual capacity) and to perform deep inspirations against the external load. The first week, the resistance will be fixed at 30% of the baseline measured maximal inspiratory pressure (MIP). Participants will be instructed to increase the resistance by 10% of the baseline set resistance each week.
  Arms: IMT
Device: EMT — A pressure threshold loading device will be used: the POWERbreathe Ex1 EMT Medic (load range 10-90 cmH2O) or POWERbreathe Ex1 EMT MR (load range 35-175 cmH2O) depending on their baseline MEP measurement. Participants will be instructed to inhale quietly during normal tidal breathing through the training device and to perform rapid and deep exhalation against the external load. The first week, the resistance will be fixed at 30% of the baseline measured MEP. Participants will be instructed to increase the resistance by 10% of the baseline set resistance each week.
  Arms: EMT
Device: Sham — A pressure threshold loading device will be used: the POWERbreathe Ex1 EMT Medic or MR, but with the resistance mechanism inside removed and replaced by a plastic ball. The same instructions will be given as for the EMT group, except that there will be no or minimal resistance (less than 6 cmH2O). There will be no change in resistance over the weeks.
  Arms: Sham

SUMMARY:
This study aims to investigate the effects of respiratory muscle training on tongue muscle function in healthy subjects. We hypothesize that respiratory muscle training can improve strength and endurance of the tongue muscles.

DETAILED DESCRIPTION:
In patient with obstructive sleep apnea, studies have shown that respiratory muscle training improved sleep-related outcomes in patients with obstructive sleep apnea (OSA). On the other hand, a recent study showed that expiratory muscle training improved tongue motor strength in patients with OSA. We hypothesize that respiratory muscle training (either Inspiratory Muscle Training (IMT) or Expiratory Muscle Training (EMT)) may elicit sleep-related improvement in patient with OSA through enhancement on tongue muscle function.

To investigate our hypothesis, we will first address this question in a population of healthy subjects. This study will therefore investigate the effects of respiratory muscle training on tongue muscle function in healthy subjects. The primary hypothesis is that the IMT program with lead to an increase in tongue strength compared to the control group. Other hypothesizes are that EMT, but not sham, will also lead to an increase in tongue strength, compared to the control group.

ELIGIBILITY:
Inclusion Criteria:

Community ambulant adults between 18 to 65 years old as of testing day; able to understand French or Dutch (depending on the study's site of inclusion); BMI ≥ 18 and ≤ 30 kg/m².

Exclusion Criteria:

Any diagnosed neuromuscular or cardiorespiratory disease; diagnosed psychiatric or psychological disorders which could affect adherence to or comprehension of instructions; diagnosed eating disorders; previous or ongoing head and neck cancer; diagnosed OSA; presenting a high-risk of sleep-disordered breathing indicated by a NoSAS score of 8 or higher 32 or a STOP-Bang score of 3 or higher 33,34; resting heart rate (HR) > 100 beats per minute (bpm) or < 50 bpm; resting systolic blood pressure (SBP) > 140 or < 90 mmHg, diastolic blood pressure (DBP) > 90 or < 50 mmHg; oxygen saturation (SpO2) < 94% at rest on room air. Individuals with abnormal lung function, i.e., forced expiratory volume in 1 second (FEV1) ≤ 80%, forced vital capacity (FVC) ≤ 80%, and FEV1/FVC ≤ 70%, will also be excluded.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2024-11-04 (Actual); Primary Completion 2025-11-01 (Estimated); Study Completion 2026-03-01 (Estimated)

PRIMARY OUTCOMES:
Tongue elevation strength | Measured two times: at baseline and after 8 weeks
  Tongue elevation strength (peak pressure) will be measured via the Iowa Oral Performance Instrument (IOPI).

SECONDARY OUTCOMES:
Tongue protrustion strength | Measured two times: at baseline and after 8 weeks
  Tongue protrusion strength (peak pressure) will be measured via the Iowa Oral Performance Instrument (IOPI).
Tongue elevation endurance | Measured two times: at baseline and after 8 weeks
  Tongue elevation endurance (50% of peak pressure) will be measured via the Iowa Oral Performance Instrument (IOPI).
Tongue protrusion endurance | Measured two times: at baseline and after 8 weeks
  Tongue protrusion endurance (50% of peak pressure) will be measured via the Iowa Oral Performance Instrument (IOPI).
Maximal inspiratory pressure | Measured two times: at baseline and after 8 weeks
  Maximal inspiratory pressure will be measured at functional residual capacity (FRC)
Maximal expiratory pressure | Measured two times: at baseline and after 8 weeks
  Maximal expiratory pressure will be measured at total lung capacity (TLC)
Snoring intensity | Measured two times: at baseline and after 8 weeks
  The participants' bed partners (if applicable) will be asked to rate their partner´s snoring using a Visual Analog Scale (VAS), which ranked the impact of snoring from 0 (no snoring) to 10 (intolerable).
Tongue base thickness | Measured two times: at baseline and after 8 weeks
  This measurement will be performed with a portable ultrasound machine
Total sagittal thickness | Measured two times: at baseline and after 8 weeks
  This measurement will be performed with a portable ultrasound machine
Lateral pharyngeal wall thickness | Measured two times: at baseline and after 8 weeks
  This measurement will be performed with a portable ultrasound machine
Snoring duration | Measured two times: at baseline and after 8 weeks
  This recording will be conducted using the standard microphone application installed on the participant's personal phone and through the use of the free, already validated in studies, SnoreLab application.

CONTACTS AND LOCATIONS:
Locations (3):
- Belgium (2):
  - KULeuven, Leuven
  - UCLouvain, Louvain-la-Neuve
- HESAV, Lausanne, Switzerland

IPD SHARING:
Plan to Share IPD: No